CLINICAL TRIAL: NCT06101147
Title: Effect of Vitamin D Supplementation on Testosterone Level in Women With Polycystic Ovary Syndrome: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Vitamin D Supplementation on Testosterone Level in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Nilufar Yasmin, Resident, MD, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BSMMU/2023/11021
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: PCOS; Vitamin D
Keywords: PCOS, Vitamin D, Testosterone
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental)
  Interventions: Drug: Vitamin D3
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Vitamin D3 — These patients will receive Vitamin D3 1000 I.U daily and the Metformin as prescribed by the physician for 8 weeks.
  Arms: Vitamin D group
Drug: Placebo Oral Tablet — These patients will receive placebo and the Metformin as prescribed by the physician for the same periods of study group
  Arms: Placebo group

SUMMARY:
The goal of this randomized, double blind, placebo-controlled clinical trial is to learn about, the effect of low dose vitamin D supplementation compares with placebo-controlled group on testosterone level in women with polycystic ovary syndrome. Half of Participants will receive vitamin D and metformin while other half placebo and metformin.

DETAILED DESCRIPTION:
PCOS poses a significant challenge to women's health and quality of life. PCOS is a common heterogenous endocrine disorder in reproductive-aged women. PCOS is characterized by the presence of polycystic ovaries, menstrual dysfunction, infertility and biochemical (elevated androgens) and clinical (hirsutism and/or acne) hyperandrogenism. Hyperandrogenism and insulin resistance exacerbate one another in the development of PCOS, Research has suggested a potential link between Vitamin D deficiency and the prevalence and severity of PCOS. There is also evidence that Vitamin D has a direct effect on the ovaries and adrenal glands, which are the primary sites of androgen production in women. Vitamin D has been found to inhibit the synthesis of androgens in these glands, suggesting that it could potentially be used to manage hyperandrogenism in women with PCOS. Furthermore, studies have shown that Vitamin D supplementation can reduce insulin resistance in women with PCOS, which can subsequently lead to a decrease in the overproduction of androgens. may improves menstrual irregularities.

In human ovarian tissue, vitamin D stimulation of oestrogen and progesterone production and lack of effect on testosterone production may be explained by the expression of the aromatase gene and augmentation of aromatase activity by vitamin D.

Serum 25OH-D level has been shown to be negatively correlated with serum androgen levels DHEAS, testosterone and hirsutism. Assumption that vitamin D supplementation may also have a positive impact on serum testosterone levels. Metformin is prescribed for reducing IR in PCOS women. This is a double-blind, randomized placebo-controlled trial in PCOS women who are receiving Metformin therapy. The intervention group will receive Vitamin D Cholecalciferol (D3) 1000 I.U daily for 8 weeks, with the Metformin as prescribed by the physician whereas control group will receive placebo with Metformin during the study period. We will compare change of Total Testosterone, Vitamin D level, Fasting blood glucose, Hirsutism, Menstrual regularities and BMI, at the time of recruitment with after 8 weeks intervention in both the intervention and placebo controlled groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed case of PCOS

Age 18 years to 45 years

Exclusion Criteria:

* Pregnancy, lactating women

Diagnosed case of diabetes mellitus, liver disease, heart disease, kidney stones and disease, Tuberculosis, hyperparathyroidism

Patients receiving vitamin D, calcium supplementation within the last two months

Known hypersensitivity to Vitamin D

Patients unwilling to participate or unwilling to give written consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Total Testosterone | 1 year
  The estimated testosterone level, is 15-46 ng/dL for a reproductive aged normal menstrual cycles woman . The results demonstrate that there is a diurnal rhythm of testosterone secretion during in girls, with the highest levels in the morning 6 am-10 am .Biochemical hyperandrogenism (TT >46 ng/dl)

SECONDARY OUTCOMES:
Fasting blood glucose | 1 year
  Impaired fasting glucose (IFG) when FBG is between 5.6-6.9 mmol/L
Menstrual regularity | 1 year
  * Polymenorrheic (<21 days),
  * Eumenorrheic (21 - 35 days),
  * Oligomenorrheic (36 days - 3 months) and
  * Amenorrheic (>3 months)
Hirsutism | 1 year
  mFG score of ≥6
Vitamin D | 1 Year
  A blood level of less than 20 ng/ml is considered deficiency, insufficiency is 21- 29 ng/ml, and sufficiency is 30 ng/ml or higher.
BMI | 1 Year
  Status BMI Underweight 15-19.9 Normal weight 20-24.9 Overweight 25-29.9 Class I Obesity 30-34.9 Class II Obesity 35-39.9 Class III Obesity ≥ 40

CONTACTS AND LOCATIONS:
Overall Officials: Nilufar Yasmin, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes